CLINICAL TRIAL: NCT03649958
Title: Randomized Controlled Trials of Closed-loop Allostatic Neurotechnology to Improve Sensory Function and Pain Management After Traumatic Brain Injury
Brief Title: Neurotechnology Following Traumatic Brain Injury
Acronym: Cereset
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brain State Technologies, LLC (Industry)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-83-8754; W81XWH1720057 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Post-Concussion Symptoms; Insomnia; Pain, Chronic; Depressive Symptoms
Keywords: concussion; mTBI; headache; insomnia; PTS; anxiety; pain; depression; sleep
MeSH Terms: conditions — Post-Concussion Syndrome; Sleep Initiation and Maintenance Disorders; Chronic Pain; Depression; Brain Concussion; Headache; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Masking Description: Study I - Single-blind (participants and outcomes assessors blinded, but technologists are not), up to 126 enrolled (target of 106 being randomized)
  Study II - Controlled (participants randomly assigned to one of two interventional arms, no blinding due to 5 or 10 sessions), up to 110 enrolled (target of 86 being randomized)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- HIRREM-SOP or Cereset (Active Comparator): HIRREM-SOP is a novel, noninvasive, closed-loop, BrainEcho, acoustic stimulation neurotechnology to support relaxation and auto-calibration of neural oscillations, using auditory tones to reflect brain frequencies in near real time. This group will have 10 sessions.
  Interventions: Device: HIRREM-SOP or Cereset
- Cereset 2x (Active Comparator): Participants randomized to the Cereset 2x group will be seated in a comfortable zero-gravity chair identical to those in the HIRREM-SOP arm. They will listen to a pattern of musical notes linked to their brain activity patterns, but also receive intermittent very low level electrical stimulation of the scalp linked to brain activity. This group will only have 5 sessions,
  Interventions: Device: Cereset 2x

INTERVENTIONS:
Device: HIRREM-SOP or Cereset — HIRREM-SOP for ten 90 minute sessions
  Arms: HIRREM-SOP or Cereset
Device: Cereset 2x — Cereset 2x for five 90 minute sessions
  Arms: Cereset 2x

SUMMARY:
This two-part study seeks to improve symptoms such as pain and sleep problems after concussion, or mild traumatic brain injury (mTBI).

Study I evaluates symptoms of mTBI through a series of 10 office sessions in which musical tones are echoed, or mirrored back in real time, to reflect one's own brain activity. Those who take part in the study will be randomly assigned to receive either tones that are based on their brain activity/brainwaves, or random tones.

Study II evaluates symptoms of mTBI through either 10 office sessions of the same acoustic stimulation linked to brain activity/brainwaves as Study I compared to 5 office sessions of acoustic stimulation plus intermittent very low level electrical stimulation of the scalp linked to brain activity.

DETAILED DESCRIPTION:
Persistent symptoms after concussion or mild traumatic brain injury (mTBI), such as pain and sleep difficulties, may be related to altered patterns of brain electrical activity, including changes in amplitude and frequency. The purpose of these two studies is to evaluate a noninvasive, closed-loop, acoustic stimulation neurotechnology, High resolution, relational, resonance-based, electroencephalic mirroring, with standard operating procedures, HIRREM-SOP. This intervention is intended to improve symptoms by supporting self-optimization of brain electrical activity. Put more simply, musical tones will be played to echo, or mirror one's own brainwaves, in real time, allowing opportunity for auto-calibration, self-adjustment, and equilibration of that brain activity. The hypothesis is that over the course of ten 90-minute sessions, symptoms related to mTBI, will improve much more with musical tones linked to brainwaves than with random tones.

Participants will be enrolled at Uniformed Services University/Walter Reed National Military Medical Center in Bethesda, MD, and Womack Army Medical Center, Fort Bragg, NC.

The 106 participants in the first part of the study can be active duty or recently retired service members, or their family members, who have had a mTBI at least three months and not more than ten years ago, with related symptoms. Participants will be randomized to either musical tones that reflect their own brain activity, or random tones. A technologist will oversee each session in which the tones are presented. Participants and those analyzing outcomes will be blinded to the nature of the acoustic stimuli received. The primary outcome will be the change in Neurobehavioral Symptom Inventory scores at three months, and the final follow-up will occur be at six months. Changes in sleep, pain, dizziness, and general quality of life will also be measured.

Study II will recruit up to 100 participants with the goal of randomizing 86 participants to one of the two interventional arms equally across the same locations with the same inclusions criteria. This study seeks to establish a non-inferiority for the shorter course intervention. The primary outcome measure will continue to be the NSI score measured post-intervention and at 3-months. Changes in sleep, pain, dizziness, and general quality of life will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* 1 Must have symptoms related to concussion or TBI, not healthy controls Age 18 years or older.
* 2 Active duty or retired military service member, or dependent beneficiary.
* 3 History of mild TBI, confirmed by administration of the Ohio State University TBI
* Identification Method Interview.
* 4 At least three months, and no more than ten years, since their most recent TBI.
* 5 Persistent symptoms temporally related, or otherwise attributable to, the TBI, such as
* headache or chronic pain, sensory disturbance including auditory, visual or other sensory
* symptoms, balance difficulties, or dizziness. After obtaining informed consent, sufficient
* severity of symptoms for entry into the study will be confirmed by administration of the
* Neurobehavioral Symptom Inventory (NSI), with a score of 23 or higher required for
* inclusion.
* 6 Willingness to be randomly assigned to one of the two treatment groups and to provide
* data for all study measures.
* 7 Willingness to abstain from alcohol or recreational drug use throughout the intervention
* period and up to 3 weeks after completion of the final office-based intervention session.
* This abstention period is intended to support the stabilization of new brain activity
* patterns that may result from the intervention.
* 8 For individuals using any of the following medication classes (either regularly scheduled
* or PRN), a willingness both to discontinue or hold those medications at least five (5) halflives
* prior to the initiation of study procedures, and throughout the period of participation
* in the study, as well as to sign a release enabling contact between study staff and their
* prescribing provider, to ensure that the prescriber deems that holding said medication
* during the study period is permissible and reasonable: benzodiazepines, opioids, antipsychotics,
* mood-stabilizers, anti-convulsants, non-benzodiazepine sleep aids (including
* but not limited zolpidem, eszoplicone, zaleplon, trazadone, and diphenhydramine), other
* prescribed sedative-hypnotics, or medical marijuana or cannabinoid medication.
* 9 Willingness to abstain from initiation of PRN/as needed usage of the above listed
* medications throughout the period of study participation. This criterion only applies to
* new PRN prescription or usage. There is no requirement to abstain from a new, regularly scheduled prescription for one of the above medications during the course of the study, if the participant's provider
* deems such usage to be indicated. The potential impact of the initiation of any such
* medications during the study will be assessed by conducting sensitivity analyses after the
* completion of the study.
* 10 Willingness to alert study investigators of any changes in their medication usage
* throughout the course of their study participation.

Exclusion Criteria:

* 1 Unable or unwilling to demonstrate an understanding of the nature and intent of the
* study, and/or to complete informed consent procedures.
* 2 A history of moderate or severe TBI.
* 3 The diagnosis of a psychotic disorder (including schizophrenia and schizoaffective
* disorder), severe depression (PHQ-9 score > 20), bipolar disorder, or active suicidal or
* homicidal ideation.
* 4 Physically unable to come to the study visits, or to sit in a chair for up to two hours.
* 5 Inability to hear and repeat a phrase spoken at normal conversational volume.
* 6 Meeting criteria for a current alcohol or substance use disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory (NSI) | decrease in the score three months following enrollment
  0 = None - Rarely if ever present; not a problem at all and 4= Very Severe - Almost always present and I have been unable to perform at work, school or home due to this problem; I probably cannot function without help.

SECONDARY OUTCOMES:
PATIENT'S GLOBAL IMPRESSION OF CHANGE (PGIC) SCALE | Score increases three months after enrollment
  * No change (or condition has gotten worse) (1); to
  * A great deal better and a considerable improvement that has made all the difference (7)
HIT-6 Headache Impact Test | improve headache patterns by decreasing point score 3 months after enrollment
  based on scale from never (6 pts) to always (13 pts)
The Dizziness Handicap Inventory ( DHI ) | Lower the point total for those whose base line is greater than 10 pts at evaluation 3 months following enrollment
  To each item, the following scores can be assigned:
  No=0 Sometimes=2 Yes=4
  Scores:
  Scores greater than 10 points should be referred to balance specialists for further evaluation.
  16-34 Points (mild handicap) 36-52 Points (moderate handicap) 54+ Points (severe handicap) Scores are assigned No=0 Sometimes=2 Yes=4; total greater than 10 requires further evaluation and 54+ severe handicap
PCL-5 The PTSD Checklist for DSM-5 | Lower the score three months after enrollment
  Questions scored as 0=not at all; to, 4=Extremely
Patient Health Questionnaire-9 (PHQ-9) | Lower the score three months after enrollment
  Frequency of being bothered by the conditions where 0=not at all; to 3=nearly every day

OTHER OUTCOMES:
Defense and Veterans Pain Rating Scale | Score decrease three months after enrollment
  (0) No Pain; to (10) As bad as it could be nothing else matters.
Insomnia Severity Index | Score decrease three months after enrollment
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Automated Neuropsychological Assessment Metrics (ANAM) | improve reaction times three months after enrollment
  used to measure simple reaction time and procedural reaction time

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Uniformed Services University, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tegeler CL, Haight TJ, Cole WR, Shaltout HA, Choi YS, Harris TE, Rachels N, Bellini PG, Roy MJ, Tegeler CH. Acoustic neuromodulation with or without micro-voltage tACS reduces post-concussive symptoms. Brain Inj. 2025 May 12;39(6):496-508. doi: 10.1080/02699052.2024.2445709. Epub 2025 Feb 6. PMID 39913294
- [Derived] Cole WR, Tegeler CL, Choi YS, Harris TE, Rachels N, Bellini PG, Haight TJ, Gerdes L, Tegeler CH, Roy MJ. Randomized, controlled clinical trial of acoustic stimulation to reduce postconcussive symptoms. Ann Clin Transl Neurol. 2024 Jan;11(1):105-120. doi: 10.1002/acn3.51937. Epub 2023 Nov 22. PMID 37990636